CLINICAL TRIAL: NCT02578485
Title: Single Session of Active Video Game Promotes Post Exercise Hypotension in Middle-aged Hypertensive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Taís Feitosa da Silva, Post-graduate, Federal University of Paraíba
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: FUParana
Record Dates: First submitted 2015-10-10; First posted 2015-10-19 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- AVideogame (Experimental): Session with active video game lasting 60 minutes performing heart rate measurements every 10 minutes and evaluating the perceived exertion.
  Interventions: Device: AVideogame
- SVideogame (Active Comparator): Session with active video sedentary lasting 60 minutes performing heart rate measurements every 10 minutes and evaluating the perceived exertion.
  Interventions: Device: SVideogame
- EMIntensity (Placebo Comparator): Session with walk on a treadmill with moderate intensity lasting 60 minutes performing heart rate measurements every 10 minutes and evaluating the perceived exertion.
  Interventions: Device: EMIntensity
- EISVideogame (Placebo Comparator): Session with walk on a treadmill with intensity similar reached in session with VGA and lasting 60 minutes performing heart rate and perceived exertion measurements every 10 minutes.
  Interventions: Device: EISVideogame
- Control (Sham Comparator): Participants remained for 60 minutes at rest performing heart rate measurements every 10 minutes and evaluating the perceived exertion.
  Interventions: Device: Control

INTERVENTIONS:
Device: AVideogame — Participants active video game played by a period of 60 minutes, then remain at rest for the evaluation of post-exercise blood pressure for an additional period of 60 minutes.
  Arms: AVideogame
Device: SVideogame — Participants sedentary video game played by a period of 60 minutes, then remain at rest for the evaluation of post-exercise blood pressure for an additional period of 60 minutes.
  Arms: SVideogame
Device: EMIntensity — Participants performed walking on a treadmill at moderate intensity by a period of 60 minutes, then remain at rest for the evaluation of post-exercise blood pressure for an additional period of 60 minutes.
  Arms: EMIntensity
Device: EISVideogame — Participants performed walking on a treadmill in intensity similar to the game by a period of 60 minutes, then remain at rest for the evaluation of post-exercise blood pressure for an additional period of 60 minutes.
  Arms: EISVideogame
Device: Control — participants remained at rest for a period of 60 minutes, then remain at rest for the evaluation of post-exercise blood pressure for an additional period of 60 minutes.
  Arms: Control

SUMMARY:
Background: The active video game (VGA) it has been studied how much to the physiological factors of your practice. The objective was to determine whether an AVG session promotes post-exercise hypotension (PEH) similar to walking exercise. Methods: Fifteen hypertensive (49.0 ± 1.6 years), both genders performed five randomized sessions, lasting 60 minutes: 1) AVG, 2) sedentary video game (SVG), 3) walk treadmill with moderate intensity (WMI), 4) walk treadmill with similar intensity to VGA (WGI), and 5) control without exercise (CON). Intensity was determined by Heart rate (HR) and Perceived Exertion (PE). Blood pressure (BP) and cardiac autonomic modulation (CAM) measurements were taken at rest and every 10 minutes post exercise for 60 minutes.

DETAILED DESCRIPTION:
Volunteers of study Participated of this study 15 hypertensive patients of both genders, five of them men. All participants were obese grade I and were using drug therapy. Were adopted as inclusion criteria: 1) be hypertensive; 2) age between 45 and 59 years old and 3) not perform regular exercise; 4) not use of beta-blockers drugs and calcium channel blockers; 5) not be affected by labyrinthitis; 6) women be not in menopause, and, 4) be not practitioners of VGA. Already as exclusion criteria: 1) modifying the antihypertensive treatment during treatment; and 2) Not have developed the ability to play during the adaptation period.

This study was approved by the Ethics in Research Committee of the University Hospital Lauro Wanderley under protocol nº 201/11 and after subjects having been cleared up all the procedures of the study, the subjects were asked to sign the Term of Free and Informed Consent (TFIC) according to the Resolution 196/96 of the National Health Council.

Study Design The subjects were submitted to five protocols lasting 60 minutes: 1- Game in VGA (Dance Dance Revolution ®); 2- Walking/running reproducing the intensity obtained in the session with VGA; 3- Walking/running with intensity between 60% and 85% of MHR; 4- sedentary video game (VGS) and 5- A session control without exercise (CON), where participants remained at rest. The order of sessions was determined randomly and were carried at with a minimum of 48 hours between them. The intensity was monitored by measurements of HR and PE. BP and cardiac autonomic modulation (CAM) were assessed before and for a period of 60 minutes after exercise, at intervals of 10 minutes between each measurement.

Adaptation to the game and instructions before study Before starting the experimental protocols, the volunteers performed three sessions of adaptation with 20 minutes duration each. In these sessions, they were instructed about the proper way of handling the VGA and VGS instruments, which were passed the necessary guidance on the different directions of arrows used in the game. These three sessions proved sufficient for them to understand the dynamics of the two games and obtain enough coordination to play without interruption.

After adaptation period, a schedule was made with voluntaries to the experimental procedures and they were instructed not to drink caffeine-containing foods and drinking alcoholic beverages for at least 48 hours before of the each experimental session.

AVG and SVG procedures The VGA utilized was Dance Dance Revolution® (SSD Company Ltd., Shiga, Japan) to Playstation 2® (San Mateo, CA, USA). In this VGA the practitioner simulates a synchronized dance for footsteps ordered on a carpet (matpad) containing the areas to be trodden that replace traditional buttons of a control VGS. The style of the music used in the game is similar to those used in gyms. The game consists of passing arrows in four directions that appears on the screen at randomly and in the rhythm of different songs contained in the game. When the arrows pass on the screen, the player must step on the corresponding arrow on the carpet, in the music rhythm. At the end of each music, immediately next music was selected to minimize the time interval between them. Was connected to the video game a multimedia projector used as screen, where it was played the game image.

The VGS game was the same as VGA, with the difference only that the carpet was replaced by joystick and volunteers remained seated during the game. Both sessions VGA as VGS lasted for 60 minutes. Heart rate was measured every 10 min using um heart rate monitor (Polar ® brand, model RS800CX, Polar ElectroOy, Kempele, Finland).

Aerobic Exercise Protocol The subjects performed two aerobic exercise sessions lasting 60 minutes on a treadmill (Moviment® LX160i - Brudden LTDA, Amazon, Brazil). One session was performed in intensity similar to the intensity reached during the session VGA and the other session was performed with moderate intensity (ranged between 60% to 85% of maximum reserve heart rate).

Heart rate was monitored by heart rate monitor (Polar ® brand, model RS800CX, Polar ElectroOy, Kempele, Finland) every 10 minutes to ensure that volunteers maintain the predetermined intensity during exercise on treadmill. For the exercise protocol on the treadmill in the intensity of AVG, the lowest and highest measured heart rate found in the video game was adopted as a target zone for the heart rate on the treadmill. To the protocol on moderate intensity, the target heart rate was determined according to equation (equation 1) proposed by Karvonen, et al.20:

Equation I FCT = FCR + i%(FCM-FCR), FCT= heart rate training; FCR = heart rate at rest;; FCM = Maximum heart rate; i% = training intensity

During the rest period the Subjective Perception Scale of Borg effort 21 was presented to the subjects with indices 6-20 for the subjects become acquainted with fatigue stages that are from very mild to exhaustive. During the games or exercise on the treadmill, the PE was questioned every 10 minutes.

Blood Pressure Monitoring After the arrival of the subjects to the data collection site, they were instructed to remain seated for 10 minutes in a quiet room, illuminated with controlled temperature between 295,1ºC and 298,1ºC and then was measured the baseline BP. New BP measurements were taken immediately after the end of exercise and for 60 minutes of the post exercise or video game procedures recovery every 10 minutes. BP was measured by auscultation, following strictly the protocol proposed in the VI Brazilian Guidelines on Hypertension22. For Was used a aneroid sphygmomanometer (WelkinAlllyn®, Skaneateles Falls, New York, USA) with an accuracy of two millimeters of mercury and previously calibrated against a mercury column and a stethoscope Premiun® mark (G-Tech).

Cardiac Autonomic Modulation (CAM) CAM was determined by recording the variability RR interval of HR, using the hear rate monitor Polar ® RS800CX (Polar ElectroOy, Kempele, Finland). The CAM was recorded after 10 minutes of initial rest and recovery post treadmill or video game procedures for 60 minutes every 10 minutes. Each measure lasted five minutes. Data were transported through an infrared device to a computer provided with software of the same manufacturer. The data are analyzed in the frequency domain (sympathetic-vagal balance - LF / HF) in software Kubios (University of Eastern Finland, Kuopio, Finland).

ELIGIBILITY:
Inclusion Criteria:

1. be hypertensive;
2. age between 45 and 59 years old;
3. not perform regular exercise;
4. not use of beta-blockers drugs and calcium channel blockers;
5. not be affected by labyrinthitis
6. women be not in menopause;
7. be not practitioners of VGA.

Exclusion Criteria:

1. modifying the antihypertensive treatment during treatment;
2. Not have developed the ability to play during the adaptation period.

Ages: 45 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Change from baseline Bood Pressure at 60 minutes post exercise in the same experimental session